CLINICAL TRIAL: NCT06010901
Title: A Phase Ib Clinical Study to Evaluate the Efficacy and Safety of of TQB2618 Injection Monotherapy and Combination Regimen (With Penpulimab Injection ±Anlotinib Hydrochloride Capsules) in the Four or Later Lines of Treatment of Advanced Colorectal Cancer.
Brief Title: A Clinical Study of TQB2618 Injection Monotherapy and Combination Regimen (With Penpulimab Injection ±Anlotinib Hydrochloride Capsules) in the Four or Later Lines of Treatment of Advanced Colorectal Cancer.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQ2618-AK105-Ib-05
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2023-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — penpulimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TQB2618 injection+Penpulimab injection +Anlotinib hydrochloride capsules (Experimental): TQB2618 injection combined with Penpulimab injection and Anlotinib hydrochloride capsules, 3 weeks as a treatment cycle.
  Interventions: Drug: TQB2618 injection; Drug: Penpulimab injection; Drug: Anlotinib hydrochloride capsules
- TQB2618 injection+Penpulimab injection (Experimental): TQB2618 injection combined with Penpulimab injection, 3 weeks as a treatment cycle.
  Interventions: Drug: TQB2618 injection; Drug: Penpulimab injection
- TQB2618 injection (Experimental): TQB2618 injection, 3 weeks as a treatment cycle.
  Interventions: Drug: TQB2618 injection

INTERVENTIONS:
Drug: TQB2618 injection — TQB2618 is a monoclonal antibody targeting T cell immunoglobulin and mucin domain-3 (TIM-3) receptor.
Drug: Penpulimab injection — Penpulimab is a humanized Immunoglobulin G-1 (IgG1) monoclonal antibody that binds to human programmed cell death 1 (PD-1), a cell membrane protein that is primarily expressed on activated T cells and inhibits T cell activation.
  Arms: TQB2618 injection+Penpulimab injection; TQB2618 injection+Penpulimab injection +Anlotinib hydrochloride capsules
Drug: Anlotinib hydrochloride capsules — Anlotinib hydrochloride is a muti-target tyrosine kinase inhibitor.
  Arms: TQB2618 injection+Penpulimab injection +Anlotinib hydrochloride capsules

SUMMARY:
This is a Phase Ib clinical study to evaluate the efficacy and safety of TQB2618 injection as monotherapy and a combination regimen (with Penpulimab injection ± Anlotinib hydrochloride capsules) in the treatment of advanced colorectal cancer. 75 participants will be enrolled in the study. Objective response rate (ORR) as assessed by Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1 is the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years old; Eastern Cooperative Oncology Group Performance Status (ECOG PS) score: 0-1; Expected survival of more than 3 months;
* Histologically/cytologically confirmed metastatic colorectal cancer;
* The subjects should provide tumor tissues that meet the requirements for mismatch repair protein detection and Programmed cell death-Ligand 1 (PD-L1) expression level detection;
* Advanced colorectal cancer that progresses or is intolerant after receiving ≥3 lines of standard therapy;
* Failure of treatment with at least one of these drugs (TAS-102, Regorafenib, Fruquintinib);
* Confirmed presence of at least one measurable lesion according to Response Evaluation Criteria In Solid Tumors 1.1 (RECIST 1.1) criteria;
* Body weight ≥40 kg and Body Mass Index (BMI) ≥18.5 kg/m^2.
* The function of the main organs is good, and the laboratory examination meets the requirements;
* Female subjects of reproductive age should agree to use contraception during the study period and for 6 months after the end of the study; Male subjects should agree that contraception must be used during the study period and for 6 months after the end of the study period.

Exclusion Criteria:

* Have had or are currently suffering from other malignant tumors within 3 years;
* Have any poorly controlled cardiovascular clinical symptoms or diseases;
* Patients with ulcerative colitis and Crohn's disease; Patients with active inflammatory bowel disease within the first 4 weeks of enrollment;
* Symptoms of hematemesis and hematochezia occurred within 6 months before screening, and the daily bleeding volume ≥ 2.5 mL;
* The presence of unmitigated toxic reactions of grade 1 or above as assessed per Common Terminology Criteria for Adverse Events (CTC-AE) due to any treatment prior to first administration, excluding hair loss;
* Patients who had received Programmed Death 1 (PD-1) or PD-L1 monoclonal antibody treatment and experienced ≥ grade 3 immune-related adverse reactions or stopped immune checkpoint inhibitor treatment due to immune-related adverse reactions;
* Active or uncontrolled severe infection (≥CTC AE grade 2 infection);
* Decompensated cirrhosis, active hepatitis;
* Poor diabetes control (fasting blood glucose > 10 mmol/L);
* Patients with renal failure requiring hemodialysis or peritoneal dialysis;
* Have a clear history of neurological or psychiatric disorders, including epilepsy or dementia, and require treatment;
* Had undergone a major surgical, open biopsy or significant traumatic injury within 4 weeks prior to the first dose of the study or expected to require major surgery during the study treatment.
* Patients with arterial/venous thrombosis events, such as cerebrovascular accident, deep vein thrombosis and pulmonary embolism, occurred within 6 months before the study treatment;
* Ascites with clinical significance, including any ascites that can be found by physical examination, ascites that have been treated in the past or still need to be treated, and only those who show a small amount of ascites but no symptoms on imaging can be included; Patients with an equal or greater amount of fluid in both pleural cavities, or a large amount of fluid in one pleural cavity, or have caused respiratory dysfunction and need drainage;
* The presence of unhealed wounds, ulcers or fractures;
* Have active tuberculosis, or have a history of active tuberculosis infection within 1 year prior to enrollment, or have a history of active tuberculosis infection more than 1 year prior to enrollment, but are not receiving treatment;
* There is a history of idiopathic pulmonary fibrosis, institutional pneumonia, drug-induced pneumonia, radiation pneumonia requiring treatment or active pneumonia with clinical symptoms, and interstitial lung disease requiring steroid hormone therapy;
* Have a history of immunodeficiency, including Human Immunodeficiency Virus (HIV) positive or other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation or hematopoietic stem cell transplantation;
* Imaging shows that the tumor has invaded large blood vessels or is not clearly demarcated with blood vessels;
* Known central nervous system metastatic and/or cancerous meningitis;
* Have multiple factors that affect oral medication (such as inability to swallow, chronic diarrhea, and intestinal obstruction);
* Allergic to the ingredients of the investigational pharmaceutical preparations or excipients, or allergic to similar drugs;
* An active autoimmune disease requiring systemic treatment (e.g., disease-modifying drugs, corticosteroids, or immunosuppressants) has occurred within 2 years prior to initial medication;
* Have been diagnosed with immune deficiency or are receiving systemic glucocorticoid therapy or any other form of immunosuppressive therapy (dose > 10 mg/day prednisone or other therapeutic hormone) and continue to use within 2 weeks before the first dose;
* History of live attenuated vaccine vaccination within 28 days before the first dose or planned live attenuated vaccine vaccination during the study period;
* Have received systematic anti-tumor therapy and other interventional anti-tumor drug clinical trials such as radical surgery, chemotherapy, radical radiotherapy or immunotherapy, biotherapy, etc. within 4 weeks before the start of the study treatment;
* Within 2 weeks prior to the first drug use, the treatment of Chinese patent drugs with anti-tumor indications specified in the National Medical Products Administration (NMPA) approved drug instructions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-01-13 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | From first administration until disease progression or withdrawal due to other reasons, estimated to not exceed 8 months.
  According to RECIST 1.1 or Modified RECIST 1.1 for immune based therapeutics, (iRECIST) criteria, the proportion of subjects whose confirmed tumor volume reduction reached the pre-specified value and maintained the minimum time-frame requirements, i.e., the proportion of subjects with complete response (CR) and partial response (PR).

SECONDARY OUTCOMES:
Overall survival (OS) | Baseline up to death, estimated to not exceed 12 months
  The time from randomization to death from any cause.
Progress free survival (PFS) | From randomization to the time of disease progression or death from any cause, estimated to not exceed 12 months.
  The time from randomization to the first disease progression or death from any cause, whichever occurs first.
Disease control rate (DCR) | From first administration to the time of disease progression or withdrawal from any cause, estimated to not exceed 12 months.
  Percentage of subjects with complete response, partial response, or stable disease as determined by RECIST 1.1 or iRECIST.
Duration of response (DOR) | From first administration to the time of disease progression or death from any cause, estimated to not exceed 12 months.
  From the time the tumor first assessed as complete or partial response to the time of first disease progression or death from any causes.
The incidence of adverse event (AE) | From first administration to 28 days after withdrawal or the start time of the new anti-tumor treatment, whichever comes first.
  The incidence and severity of adverse events as determined by the Common Terminology Criteria for Adverse Events (CTC AE).
Anti-drug antibodies (ADA) | Cycle 1 Day 1, Cycle 2 Day 1, Cycle 4 Day 1, Cycle 8 Day 1, 30 days and 90 days after the last dose. Each cycle is 21 days.
  The occurrence of ADA
Neutralizing antibodies (NaB) | Cycle 1 Day 1, Cycle 2 Day 1, Cycle 4 Day 1, Cycle 8 Day 1, 30 days and 90 days after the last dose. Each cycle is 21 days.
  The occurrence of neutralizing antibodies

CONTACTS AND LOCATIONS:
Locations (15):
- China (15):
  - Fuyang Cancer Hospital, Fuyang, Anhui
  - Huai Nan First People's Hospital, Huainan, Anhui
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Meizhou People's Hospital (Huangtang Hospital), Meizhou, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of Air Force Medical University, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Jiao Tong University, Xi'an, Shaanxi
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - The people's hospital of Leshan, Leshan, Sichuan
  - Mianyang central hospital, Mianyang, Sichuan